CLINICAL TRIAL: NCT04100200
Title: Polyphenols and Human Gut Microbiome Interactions: Role of in Ameliorating Inflammation
Brief Title: Berries, Inflammation, and Gut Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB2018-121
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Overweight or Obesity; Healthy
Keywords: Strawberry; Raspberry; Metabolic responses; Gut microbiome; Inflammatory markers
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mixed Berries (Active Comparator): Strawberry and red raspberry composite served as a frozen drink
  Interventions: Dietary Supplement: Mixed berries
- FOS (Active Comparator): Non-polyphenol, carbohydrate-based fermentable fiber/pre-biotic served as a frozen drink
  Interventions: Dietary Supplement: FOS
- Combination (Active Comparator): Mixed berry composite + FOS served as a frozen drink
  Interventions: Dietary Supplement: Combination
- Control (Placebo Comparator): Placebo similar in color to mixed berry supplement without any polyphenols served as a frozen drink
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Mixed berries — Strawberry and red raspberry
  Arms: Mixed Berries
Dietary Supplement: FOS — Fructo-oligosaccharide
  Arms: FOS
Dietary Supplement: Control — Placebo similar in color to mixed berry supplement without any polyphenols
  Arms: Control
Dietary Supplement: Combination — Mixed berry composite + FOS
  Arms: Combination

SUMMARY:
The primary objectives are to characterize changes in indices of systemic and gut inflammation, assess host- and microbial-derived metabolite pools, and describe and link functional metagenomics and metatranscriptomic alterations in the gut microbiome with metabolite and inflammatory outcomes after acute (24hr) and chronic (4 week) intake of anthocyanins and ellagitannins from strawberry and red raspberries compared to a control diet (negative control), FOS (positive control, non-polyphenol, carbohydrate-based fermentable fiber/pre-biotic), or combination diet (berry composite + FOS) in human participants with low-grade inflammation.

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening.

This is a single-center, randomized, single-blinded, 4-arm, placebo-controlled clinical trial. It features an acute single exposure 24-h protocol and a chronic 4-week daily intake protocol to evaluate the effects of anthocyanins and ellagitannins from strawberry and red raspberry intake compared to a control diet, FOS, or FOS and berries combined on gut inflammation, in adults with chronic low-grade inflammation.

A planned sample size of 88 will be enrolled in the study. This study will require one initial screening visit, a pre-study visit, and 5 study visits. This study will take 5 weeks per subject to complete.

The initial screening visit will provide subject with their site-specific, IRB-approved informed consent document prior to the start of any study-related procedures. Subject eligibility will be determined through a high sensitivity C-Reactive Protein (hs-CRP) marker value, anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey related to general eating, health, mood and exercise habits.

Eligible subjects will follow a limited polyphenolic diet throughout the duration of their participation, although stricter guidelines will be imposed during the 3 days prior to a study visit that involved blood/urine/fecal collection. Shopping lists and meal plans will be provided to subjects, along with counseling by the investigator's study investigators, to help subjects adhere to the limited polyphenolic diet. The trial will initiate with a 3-day food diary to assess background (pre-study) dietary intake followed by counseling to follow a diet relatively low in (poly)phenolic rich-beverages/foods, which will be maintained for the duration of the experiment. After an initial 7-day wash-in period on the limited polyphenolic diet, subjects will be randomized to 1 of 4 treatment sequences in the form of a drink: a mixed berries diet (raspberries and strawberries), a FOS diet (non-polyphenol, carbohydrate-based fermentable fiber/pre-biotic), a combination diet (mixed berries + FOS), or a control diet (negative control). Subjects will receive the same treatment for the duration of the study. Treatment codes will be maintained by the principal investigator.

Each visit will last ~2 hours and subjects will be required to remain at the Clinical Nutrition Research Center for the duration of the visit. Fasting blood samples will be collected at the 0 and 24h time points via a butterfly needle placed by a certified phlebotomist.

ELIGIBILITY:
Inclusion Criteria

* C-Reactive Protein (hs-CRP) > 1.0 and ≤ 10 ng/L
* BMI ≥ 25 kg/m2
* Aged 20-60 years
* Able to provide informed consent and comply with study procedures
* Willing to maintain stable body weight and follow his/her habitual diet and physical activity patterns throughout the trial.
* Judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.
* People with no documented disease condition that would interfere with the study endpoints (ie., CVD, diabetes, hypertension, major organ diseases) or taking medication or dietary supplements that may interfere with study endpoints

Exclusion Criteria

* Current smoker or marijuana user
* No history or presence of atherosclerosis/cardiovascular disease, inflammatory disease, diabetes mellitus, or other systemic diseases, psychological or psychiatric disorders that may interfere with study outcomes.
* Taking any medications and/or supplements that would interfere with outcomes of the study (i.e., lipid-lowering medications, anti-inflammatory drugs, etc)
* Take part in prebiotics, probiotics or drugs active on gastrointestinal motility or a laxative of any class within 1 month
* Unstable use of any medication/supplement, this could include marijuana used as -needed for medical reasons
* Have a history of cancer, except for non-melanoma skin cancer in past 5 years
* Addicted to drugs and/or alcohol (>4 drinks/day)
* Have been exposed to any non-registered drug product within last 30 days.
* Working overnight (e.g. 3rd shift of overnight workers)
* Excessive exercisers or trained athletes
* Have allergies/intolerances to any of the study products.
* Extreme dietary habits (ie. vegetarian/vegan)
* Excessive coffee/tea drinker (>4 cups/day)
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months)
* Donated blood within last 3 months
* Participated in a clinical trial within 1 month
* Female who is pregnant, planning to be pregnant, breastfeeding
* Any condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma biomarkers and measures of inflammation concentration: Nrf2/ NF-κB -response between 4 treatments | Baseline to 4 weeks
  Plasma biomarkers and measures of inflammation: Nrf2/ NF-κB activation in monocytes will be analyzed.
Changes in plasma biomarkers and measures of inflammation concentration-response between 4 treatments | Baseline to 4 weeks
  Inflammatory cytokines (Interleukin-6 (IL-6), High Sensitivity C-Reactive Protein (hs-CRP), Tumor Necrosis Factor-α (TNF-α)) will be measured.
Changes in plasma biomarkers and measures of inflammation concentration (GLP-2)-response between 4 treatments | Baseline to 4 weeks
  Analysis of GLP-2 will be done in plasma samples before and after chronic exposure to the study foods.

SECONDARY OUTCOMES:
Changes in gut inflammatory markers between 4 treatments. | Baseline to 4 weeks
  The concentration of calprotectin, zonulin, and IgA in fecal samples will be determined by enzyme-linked immunosorbent assay (ELISA) before and after chronic exposure to study foods.
Changes in Bile acids between 4 treatments. | Baseline to 4 weeks
  Bile acids in plasma and fecal samples will be determined using UHPLC-QQQ-MS.

OTHER OUTCOMES:
Characterize metabolite profiles (phenolic acids and urolithin derivatives) in urine and plasma. | Baseline to 4 weeks
  Polyphenolic metabolites (anthocyanin, ellagitannins and other phenolic components) will be identified and quantified in urine and plasma.Metabolites in samples will be identified and quantified using an Agilent 6550 iFunnel UHPLC-QTOF-MS and 6460 UHPLC-QQQ-MS, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Sandhu, Ph.D, Principal Investigator — Institue for Food Safety and Health/Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No